CLINICAL TRIAL: NCT01639703
Title: Diagnostic Contribution of XENETIX® CT PERFUSION in Pre-therapeutical Assessment of Hepatocellular Carcinoma
Brief Title: Hepatic Xenetix-CT Perfusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ISO-44-013
Record Dates: First submitted 2012-07-06; First posted 2012-07-13 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: CT perfusion; Hepatocellular Carcinoma; Xenetix; Contrast agent
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CT perfusion (Experimental): arm with CT perfusion
  Interventions: Drug: Xenetix-CT perfusion imaging

INTERVENTIONS:
Drug: Xenetix-CT perfusion imaging — Injection of 50 ml of Xenetix

SUMMARY:
The purpose of this study is to prospectively determine the diagnostic value of Xenetix-CT perfusion for the discrimination between well-differentiated hepatocellular carcinomas (HCC) and poorly/moderately differentiated HCC, in histo-pathologically proven HCC, and with the aim to cover the entire liver.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed for HCC and planned for surgery (lobectomy or transplantation) within a timeframe of 30 days between first imaging procedure used for the study and surgery.

Exclusion Criteria:

* Subjects who have undergone prior TACE (TransArterial Chemo Embolization), prior RFA (Radio Frequency Ablation) or prior SIRT (Selected Internal Radio Therapy) within one year before inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2012-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Alkadhi, Principal Investigator — Zurich University Hospital
Locations (5):
- AKH, Vienna, Austria
- Universitätsklinikum Erlangen, Erlangen, Germany
- South Korea (2):
  - SMC, Seoul
  - SNUH, Seoul
- Zurich University Hospital, Zurich, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 96 patients were enrolled in 4 countries: Austria, Germany, South Korea and Switzerland.
Period: Overall Study
Arm/Group | CT Perfusion
Started | 96
Completed | 84
Not Completed | 12
Not completed — Withdrawal by Subject | 5
Not completed — Other reason | 7

BASELINE CHARACTERISTICS:
Groups:
- All Included Patients: All patients included in the study.
Arm/Group | All Included Patients
Number analyzed (Participants) | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: For one patient, the gender was missing.
  Participants
    number analyzed (Participants) | 95
    Female | 22
    Male | 73
Region of Enrollment [Number; unit: participants]
  Austria | 3
  Korea, Republic of | 85
  Switzerland | 6
  Germany | 2
Severity of cirrhosis (Child-Pugh score) [Count of Participants; unit: Participants] — Child-Pugh classification of severity of liver disease is evaluated according to the degree of ascites, the plasma concentrations of bilirubin and albumin, the prothrombin time, and the degree of encephalopathy.
  * Class A: well compensated disease
  * Class B: significant functional compromised
  * Class C: decompensated disease
  For 7 patients, this score was missing.
  Participants
    Class A | 79
    Class B | 8
    Class C | 2

OUTCOME MEASURES:

1. Primary Outcome: Blood Volume (BV) According to Degree of Lesions Differentiation
Description: The mean level of each CT perfusion parameter was compared between well differentiated and moderately/poorly differentiated lesions according to WHO classification evaluated off-site.
Time Frame: Within a week from CT perfusion to surgery
Population: A total of 77 patients were analyzed for CT perfusion parameters: 38 had lesions assessed as "well differentiated", 42 had lesions assessed as "moderately/poorly differentiated" and 3 had lesions assessed as "well differentiated" and "moderately/poorly differentiated".
Measure: Mean (Standard Deviation); unit: mL/100 grams
Units Other Than Participants: lesions
Groups:
- Well Differentiated Lesions: Among the 90 lesions analyzed for CT perfusion parameters, 47 were well differentiated according to WHO classification.
- Moderately/Poorly Differentiated Lesions: Among the 90 lesions analyzed, 43 were moderately or poorly differentiated according to WHO classification.
Arm/Group | Well Differentiated Lesions | Moderately/Poorly Differentiated Lesions
Number analyzed (Participants) | 38 | 42
Number analyzed (lesions) | 47 | 43
mL/100 grams | 15.930 (6.663) | 13.958 (5.315)

2. Primary Outcome: Blood Flow (BF) According to Degree of Lesions Differentiation
Description: as for outcome 1
Time Frame: Within a week from CT perfusion to surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/100 grams/min
Units Other Than Participants: lesions
Groups:
- Well Differentiated Lesions: Among the 90 lesions analyzed, 47 were well differentiated according to WHO classification.
Arm/Group | Well Differentiated Lesions | Moderately/Poorly Differentiated Lesions
Number analyzed (Participants) | 38 | 42
Number analyzed (lesions) | 47 | 43
mL/100 grams/min | 73.042 (21.551) | 72.051 (31.792)

3. Primary Outcome: Permeability Surface (PS) According to Degree of Lesions Differentiation
Description: as for outcome 1
Time Frame: Within a week from CT perfusion to surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/100 grams/min
Units Other Than Participants: lesions
Arm/Group | Well Differentiated Lesions | Moderately/Poorly Differentiated Lesions
Number analyzed (Participants) | 38 | 42
Number analyzed (lesions) | 47 | 43
mL/100 grams/min | 26.421 (10.014) | 27.750 (9.425)

4. Secondary Outcome: Arterial Liver Perfusion (ALP) According to Degree of Lesions Differentiation
Description: as for outcome 1
Time Frame: Within a week from CT perfusion to surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min/100 mL
Units Other Than Participants: lesions
Arm/Group | Well Differentiated Lesions | Moderately/Poorly Differentiated Lesions
Number analyzed (Participants) | 38 | 42
Number analyzed (lesions) | 47 | 43
mL/min/100 mL | 43.234 (16.989) | 42.967 (16.678)

5. Secondary Outcome: Portal Venous Liver Perfusion (PVP) According to Degree of Lesions Differentiation
Description: as for outcome 1
Time Frame: Within a week from CT perfusion to surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min/100 mL
Units Other Than Participants: lesions
Arm/Group | Well Differentiated Lesions | Moderately/Poorly Differentiated Lesions
Number analyzed (Participants) | 38 | 42
Number analyzed (lesions) | 47 | 43
mL/min/100 mL | 19.492 (14.586) | 13.708 (13.207)

6. Secondary Outcome: Total Liver Perfusion (TLP) According to Degree of Lesions Differentiation
Description: The mean level of each CT perfusion parameter was compared between well differentiated and moderately/poorly differentiated lesions according to WHO classification evaluated off-site.
  TLP = ALP + PVP
Time Frame: Within a week from CT perfusion to surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min/100 mL
Units Other Than Participants: lesions
Arm/Group | Well Differentiated Lesions | Moderately/Poorly Differentiated Lesions
Number analyzed (Participants) | 38 | 42
Number analyzed (lesions) | 47 | 43
mL/min/100 mL | 62.725 (15.620) | 56.674 (20.494)

7. Secondary Outcome: Hepatic Perfusion Index (HPI) According to Degree of Lesions Differentiation
Description: as for outcome 1
Time Frame: Within a week from CT perfusion to surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Units Other Than Participants: lesions
Arm/Group | Well Differentiated Lesions | Moderately/Poorly Differentiated Lesions
Number analyzed (Participants) | 38 | 42
Number analyzed (lesions) | 47 | 43
percentage | 75.232 (18.458) | 80.834 (14.503)

8. Secondary Outcome: Blood Volume According to Immunohistochemistry Parameter (Glutamine Synthetase)
Description: Glutamine synthetase is an immunohistochemistry parameter of hepatocellular carcinoma phenotype.
  Glutamine synthetase labelling was quantified and in case of positive quantification, classified in the following categories: 1-10%, 10-50% and >50%. In case of absence of glutamine synthetase labelling, lesions were classified in the "glutamine synthetase 0%" category.
Time Frame: Within a week from CT perfusion to surgery
Population: A total of 77 patients were analyzed for CT perfusion and immunohistochemistry parameters. A patient could have several lesions in different groups: 3 patients presented at least 1 lesion in group10-50% and another lesion in group >50%; 2 patients presented at least 1 lesion in group >50% and 1 missing data; 2 patients presented missing data.
Measure: Mean (Standard Deviation); unit: mL/100 grams
Units Other Than Participants: lesions
Groups:
- Glutamine Synthetase 0%: Absence of glutamine synthetase labelling
- Glutamine Synthetase 1-10%: Quantification of glutamine synthetase labelling from 1 to 10%
- Glutamine Synthetase 10-50%: Quantification of glutamine synthetase labelling from 10 to 50%
- Glutamine Synthetase >50%: Quantification of glutamine synthetase labelling greater than 50%
Arm/Group | Glutamine Synthetase 0% | Glutamine Synthetase 1-10% | Glutamine Synthetase 10-50% | Glutamine Synthetase >50%
Number analyzed (Participants) | 6 | 0 | 15 | 57
Number analyzed (lesions) | 6 | 0 | 17 | 62
mL/100 grams | 14.994 (5.714) |  | 12.964 (5.268) | 15.551 (6.328)
Statistical Analysis 1: Comparison: Glutamine Synthetase 0% vs Glutamine Synthetase 1-10% vs Glutamine Synthetase 10-50% vs Glutamine Synthetase >50%; Multinomial logistic regression analyses were performed with each off-site CT perfusion parameters as explicative variables taken alone and each off-site immunohistochemistry categorized parameters as dependent variables; Test type: Other; p = 0.2476, Regression, Logistic; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.47 to 1.21] — Odds-ratio is the risk to move from one immunochemistry category to the below one (among 0%, 1-10%, 10-50% and >50%) considering an increase of 5 units for Blood Volume

9. Secondary Outcome: Blood Volume According to Immunohistochemistry Parameter (CD31)
Description: CD31 is an immunohistochemistry marker of microvessel density. CD31 labelling was quantified and in case of positive quantification, classified in the following categories: 1-10%, 10-50% and >50%. In case of absence of CD31 labelling, lesions were classified in the "CD31 0%" category.
Time Frame: Within a week from CT perfusion to surgery
Population: A total of 77 patients were analyzed for CT perfusion and immunohistochemistry parameters. A patient could have several lesions.
Measure: Mean (Standard Deviation); unit: mL/100 grams
Units Other Than Participants: lesions
Groups:
- CD31 0%: Absence of CD31 labelling
- CD31 1-10%: Quantification of CD31 labelling from 1 to 10%
- CD31 10-50%: Quantification of CD31 labelling from 10 to 50%
- CD31 >50%: Quantification of CD31 labelling greater than 50%
Arm/Group | CD31 0% | CD31 1-10% | CD31 10-50% | CD31 >50%
Number analyzed (Participants) | 0 | 35 | 42 | 0
Number analyzed (lesions) | 0 | 39 | 45 | 0
mL/100 grams |  | 14.708 (7.657) | 15.589 (4.561) |
Statistical Analysis 1: Comparison: CD31 0% vs CD31 1-10% vs CD31 10-50% vs CD31 >50%; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.5354, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.77 to 1.66] — [estimate comment as in outcome 8, analysis 1]

10. Secondary Outcome: Blood Flow According to Immunohistochemistry Parameter (Glutamine Synthetase)
Description: as for outcome 8
Time Frame: Within a week from CT perfusion to surgery
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mL/100 grams/min
Units Other Than Participants: lesions
Arm/Group | Glutamine Synthetase 0% | Glutamine Synthetase 1-10% | Glutamine Synthetase 10-50% | Glutamine Synthetase >50%
Number analyzed (Participants) | 6 | 0 | 15 | 57
Number analyzed (lesions) | 6 | 0 | 17 | 62
mL/100 grams/min | 79.178 (32.656) |  | 61.804 (22.087) | 74.261 (27.619)
Statistical Analysis 1: Comparison: Glutamine Synthetase 0% vs Glutamine Synthetase 1-10% vs Glutamine Synthetase 10-50% vs Glutamine Synthetase >50%; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.3487, Regression, Logistic; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.71 to 1.13] — Odds-ratio is the risk to move from one immunochemistry category to the below one (among 0%, 1-10%, 10-50% and >50%) considering an increase of 10 units for Blood Flow

11. Secondary Outcome: Blood Flow According to Immunohistochemistry Parameter (CD31)
Description: as for outcome 9
Time Frame: Within a week from CT perfusion to surgery
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mL/100 grams/min
Units Other Than Participants: lesions
Groups:
- CD31 0%: Absence of glutamine synthetase labelling
Arm/Group | CD31 0% | CD31 1-10% | CD31 10-50% | CD31 >50%
Number analyzed (Participants) | 0 | 35 | 42 | 0
Number analyzed (lesions) | 0 | 39 | 45 | 0
mL/100 grams/min |  | 70.057 (25.317) | 75.206 (28.519) |
Statistical Analysis 1: Comparison: CD31 0% vs CD31 1-10% vs CD31 10-50% vs CD31 >50%; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.4195, Regression, Logistic; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.90 to 1.29] — [estimate comment as in outcome 10, analysis 1]

12. Secondary Outcome: Permeability Surface According to Immunohistochemistry Parameter (Glutamine Synthetase)
Description: as for outcome 8
Time Frame: Within a week from CT perfusion to surgery
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mL/100 grams/min
Units Other Than Participants: lesions
Arm/Group | Glutamine Synthetase 0% | Glutamine Synthetase 1-10% | Glutamine Synthetase 10-50% | Glutamine Synthetase >50%
Number analyzed (Participants) | 6 | 0 | 15 | 57
Number analyzed (lesions) | 6 | 0 | 17 | 62
mL/100 grams/min | 28.896 (7.207) |  | 24.840 (6.769) | 27.139 (10.714)
Statistical Analysis 1: Comparison: Glutamine Synthetase 0% vs Glutamine Synthetase 1-10% vs Glutamine Synthetase 10-50% vs Glutamine Synthetase >50%; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.7127, Regression, Logistic; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.53 to 1.54] — Odds-ratio is the risk to move from one immunochemistry category to the below one (among 0%, 1-10%, 10-50% and >50%) considering an increase of 10 units for Permeability Surface

13. Secondary Outcome: Permeability Surface According to Immunohistochemistry Parameter (CD31)
Description: as for outcome 9
Time Frame: Within a week from CT perfusion to surgery
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mL/100 grams/min
Units Other Than Participants: lesions
Arm/Group | CD31 0% | CD31 1-10% | CD31 10-50% | CD31 >50%
Number analyzed (Participants) | 0 | 35 | 42 | 0
Number analyzed (lesions) | 0 | 39 | 45 | 0
mL/100 grams/min |  | 25.434 (9.721) | 28.587 (9.832) |
Statistical Analysis 1: Comparison: CD31 0% vs CD31 1-10% vs CD31 10-50% vs CD31 >50%; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.1753, Regression, Logistic; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.86 to 2.31] — [estimate comment as in outcome 12, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during and immediately after the CT perfusion examination over a 30 min follow up period.
Groups:
- Safety Set: All included patients receiving at least one injection of Xenetix, regardless of the quantity. This set was used for safety analyses.
Arm/Group | Safety Set
Serious Adverse Events (participants affected / at risk) | 0/84
Other Adverse Events (participants affected / at risk) | 4/84
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Set (N=84)
Nausea (Gastrointestinal disorders) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All written or oral papers and publications must have the joint agreement of the investigator and the sponsor.

Each investigator agrees not to publish/submit/present the results of the study main criterion involving only the patients he/she has included.

Any abstract project will be first submitted to Guerbet at least 10 working days before submission to the congress scientific committee.